CLINICAL TRIAL: NCT02771145
Title: Clinical Evaluation of the Safety and Efficacy of FID 120947A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCE293-C001
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-10

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FID 120947A (Experimental): FID 120947A contact lens disinfecting solution used with soft contact lenses (study lenses) on a daily basis for 180 days. SCL preservative solution used standard-of-care.
  Interventions: Device: FID 120947A contact lens disinfecting solution; Device: Soft contact lenses (SCL); Device: SCL preservative solution

INTERVENTIONS:
Device: FID 120947A contact lens disinfecting solution — Investigational 3% hydrogen peroxide solution that uses a platinum catalyst for neutralization and is intended for simultaneous cleaning, protein removal, disinfecting and storage of silicone hydrogel and soft contact lenses
  Other Names: Clear Care® Plus
Device: Soft contact lenses (SCL) — Commercially available soft contact lenses worn a minimum of 8 hours each day on a daily wear basis for the duration of the study (180 days). A fresh pair will be dispensed on Day 0, Day 30, Day 60, and Day 135.
  Other Names: 2-Week Acuvue®
Device: SCL preservative solution — Commercially available solution for rinsing soft contact lenses

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of FID 120947A in soft contact lens wearers of Japanese ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Successful history of silicone hydrogel or other soft contact lens wear (except for daily disposable lenses) in both eyes during the past 3 months and history of at least 5 consecutive days of successful DAILY wear in both eyes at Visit 1;
* Best spectacle corrected distance visual acuity greater than or equal to 0.8 (decimal visual acuity) in each eye;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any ocular or systemic medical condition that may, in the opinion of the Investigator, preclude safe administration of the investigational products or affect the results of this study;
* Need to wear contact lenses on an extended wear basis (ie, overnight) during the study;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Use of a daily cleaner and/or enzyme cleaner to care for lenses at least 7 days prior to Visit 1 (use of lens rewetting drops is acceptable);
* History of intolerance or hypersensitivity to any component of the investigational products;
* Unwilling or unable to abstain from use of all over-the-counter (OTC) or prescribed topical ocular medications (except for rewetting drops) within 7 days prior to Visit 1 and for the duration of the study;
* Moderate (grade 3) or severe (grade 4) corneal edema, corneal staining, injection (limbal hyperemia, bulbar conjunctival hyperemia), tarsal abnormalities, or "other" findings;
* Corneal vascularization that is mild (grade 2) or higher;
* Conjunctival or structural lid abnormalities or abnormal corneal opacities at Visit 1;
* Current or history of ocular infection, severe inflammation or disease within 6 months prior to Visit 1;
* Any systemic disease (including allergies, respiratory infections or colds) that may affect the eye or be exacerbated by use of contact lenses or contact lens solutions;
* Use of systemic medications that may contribute to adverse ocular effects unless on a stable dosing regimen for a minimum of 30 days prior to Visit 1;
* Ocular or intra-ocular surgery and/or ocular trauma within the last 12 months (excluding placement of punctal plugs);
* Participation in any investigational clinical study within 30 days of Visit 1;
* Other protocol-specified exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Group Manager, Clinical Development, Study Director — Alcon Japan, Ltd.
Locations (1):
- Contact Alcon Japan, Ltd. for Trial Locations, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 6 study centers located in Japan.
Pre-assignment Details: Of the 91 enrolled, 1 subject was exited as a screen failure prior to treatment. This reporting group includes all treated subjects (90).
Period: Overall Study
Arm/Group | FID 120947A
Started | 90
Completed | 86
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all treated subjects (Full Analysis Set).
Arm/Group | FID 120947A
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Visibly Clean Lenses at Each Visit
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered. A lens was considered visibly clean if it had nondetectable films or deposits. Both eyes contributed to the analysis.
Time Frame: Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set, with non-missing response
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | FID 120947A
Number analyzed (Participants) | 90
Number analyzed (Eyes) | 180
percentage of eyes
  Day 7 | 92.2
  Day 30: number analyzed (Participants) | 89
  Day 30: number analyzed (Eyes) | 178
  Day 30 | 88.2
  Day 60: number analyzed (Participants) | 89
  Day 60: number analyzed (Eyes) | 178
  Day 60 | 95.5
  Day 90: number analyzed (Participants) | 87
  Day 90: number analyzed (Eyes) | 174
  Day 90 | 92.5
  Day 135: number analyzed (Participants) | 84
  Day 135: number analyzed (Eyes) | 168
  Day 135 | 95.2
  Day 180: number analyzed (Participants) | 86
  Day 180: number analyzed (Eyes) | 172
  Day 180 | 95.9

2. Primary Outcome: Number of Eyes With Film Deposits on Lens by Type at Each Visit
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered. Both eyes contributed to the analysis.
Time Frame: Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Groups:
- Type II: Films or deposits visible only under special conditions, such as special illumination using an eyepiece of 7-10 times magnification
- Type III: Films or deposits readily visible on a dry lens under room lighting, with unaided eye
- Type IV: Films or deposits obvious under room lighting, with unaided eye, when the lens is wet or dry
Arm/Group | Type II | Type III | Type IV
Number analyzed (Participants) | 90 | 90 | 90
Number analyzed (Eyes) | 180 | 180 | 180
eyes
  Day 7 | 0 | 3 | 1
  Day 30 | 3 | 0 | 4
  Day 60 | 1 | 0 | 3
  Day 90 | 1 | 1 | 2
  Day 135 | 2 | 1 | 2
  Day 180 | 1 | 0 | 1

3. Primary Outcome: Number of Eyes With Crystalline Deposits on Lens by Type at Each Visit
Description: as for outcome 2
Time Frame: Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Type II | Type III | Type IV
Number analyzed (Participants) | 90 | 90 | 90
Number analyzed (Eyes) | 180 | 180 | 180
eyes
  Day 7 | 4 | 8 | 2
  Day 30 | 5 | 4 | 8
  Day 60 | 0 | 0 | 4
  Day 90 | 1 | 0 | 10
  Day 135 | 0 | 0 | 3
  Day 180 | 0 | 0 | 5

4. Primary Outcome: Percentage of Lens Area Covered by Film Deposits at Each Visit
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered. For each visit, the number analyzed represents the number of eyes with film deposits on lens, respectively.
Time Frame: Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of lens area
Units Other Than Participants: eyes
Arm/Group | FID 120947A
Number analyzed (Participants) | 90
Number analyzed (eyes) | 180
percentage of lens area
  Day 7: number analyzed (Participants) | 3
  Day 7: number analyzed (eyes) | 4
  Day 7 | 7.5 (2.89)
  Day 30: number analyzed (Participants) | 4
  Day 30: number analyzed (eyes) | 7
  Day 30 | 28.6 (14.92)
  Day 60: number analyzed (Participants) | 4
  Day 60: number analyzed (eyes) | 4
  Day 60 | 17.5 (15.00)
  Day 90: number analyzed (Participants) | 3
  Day 90: number analyzed (eyes) | 4
  Day 90 | 15.0 (10.00)
  Day 135: number analyzed (Participants) | 4
  Day 135: number analyzed (eyes) | 5
  Day 135 | 6.0 (2.24)
  Day 180: number analyzed (Participants) | 2
  Day 180: number analyzed (eyes) | 2
  Day 180 | 7.5 (3.54)

5. Primary Outcome: Percentage of Lens Area Covered by Crystalline Deposits at Each Visit
Description: as for outcome 4
Time Frame: Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of lens area
Units Other Than Participants: Eyes
Arm/Group | FID 120947A
Number analyzed (Participants) | 90
Number analyzed (Eyes) | 180
percentage of lens area
  Day 7: number analyzed (Participants) | 8
  Day 7: number analyzed (Eyes) | 14
  Day 7 | 10.4 (7.90)
  Day 30: number analyzed (Participants) | 12
  Day 30: number analyzed (Eyes) | 17
  Day 30 | 10.8 (9.65)
  Day 60: number analyzed (Participants) | 3
  Day 60: number analyzed (Eyes) | 4
  Day 60 | 8.8 (2.50)
  Day 90: number analyzed (Participants) | 6
  Day 90: number analyzed (Eyes) | 11
  Day 90 | 7.1 (3.45)
  Day 135: number analyzed (Participants) | 2
  Day 135: number analyzed (Eyes) | 3
  Day 135 | 11.7 (7.64)
  Day 180: number analyzed (Participants) | 3
  Day 180: number analyzed (Eyes) | 5
  Day 180 | 13.0 (9.75)

6. Primary Outcome: Percentage of Eyes With Change From Baseline in Contact Lens-Corrected Distance Visual Acuity (CLCDVA) by Line Change at Each Visit
Description: Distance VA was assessed for each eye individually while reading a chart distant to the participant in dimmed room illumination. VA was measured using Decimal acuity, where 1.0 (equivalent to 20/20) is considered normal distance-eyesight. A line increase indicates an improvement in VA. Both eyes contributed to the analysis
Time Frame: Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set, with non-missing response
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | ≥3 Line Increase | 2 Line Increase | 1 Line Increase | No Change | 1 Line Decrease | 2 Line Decrease | ≥3 Line Decrease
Number analyzed (Participants) | 90 | 90 | 90 | 90 | 90 | 90 | 90
Number analyzed (Eyes) | 180 | 180 | 180 | 180 | 180 | 180 | 180
percentage of eyes
  Day 7: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89 | 89 | 89
  Day 7: number analyzed (Eyes) | 178 | 178 | 178 | 178 | 178 | 178 | 178
  Day 7 | 0.6 | 0.6 | 6.2 | 90.4 | 1.7 | 0.6 | 0.0
  Day 30: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89 | 89 | 89
  Day 30: number analyzed (Eyes) | 178 | 178 | 178 | 178 | 178 | 178 | 178
  Day 30 | 1.7 | 3.4 | 7.3 | 84.8 | 2.8 | 0.0 | 0.0
  Day 60: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89 | 89 | 89
  Day 60: number analyzed (Eyes) | 178 | 178 | 178 | 178 | 178 | 178 | 178
  Day 60 | 1.7 | 3.4 | 10.7 | 79.2 | 3.9 | 1.1 | 0.0
  Day 90: number analyzed (Participants) | 87 | 87 | 87 | 87 | 87 | 87 | 87
  Day 90: number analyzed (Eyes) | 174 | 174 | 174 | 174 | 174 | 174 | 174
  Day 90 | 0.0 | 3.4 | 11.5 | 79.9 | 4.6 | 0.6 | 0.0
  Day 135: number analyzed (Participants) | 84 | 84 | 84 | 84 | 84 | 84 | 84
  Day 135: number analyzed (Eyes) | 168 | 168 | 168 | 168 | 168 | 168 | 168
  Day 135 | 1.8 | 3.0 | 8.3 | 77.4 | 8.9 | 0.6 | 0.0
  Day 180: number analyzed (Participants) | 86 | 86 | 86 | 86 | 86 | 86 | 86
  Day 180: number analyzed (Eyes) | 172 | 172 | 172 | 172 | 172 | 172 | 172
  Day 180 | 1.2 | 2.3 | 9.9 | 75.6 | 8.1 | 1.7 | 1.2

7. Primary Outcome: Average Lens Wear Time (Averaged Over the Last 3 Days) at Each Visit
Description: Subject recorded a response to the question, "Averaging over the last 3 days, how many hours per day did you wear your contact lenses?" Lens wear time was summarized as an estimate of the subject's daily wear, averaged over the course of 3 days prior to each scheduled visit, and measured in hours. Habitual lenses were used at the Day 0 time point.
Time Frame: Day 0, Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set, with non-missing response
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | FID 120947A
Number analyzed (Participants) | 90
hours
  Day 0 | 12.4 (2.54)
  Day 7 | 11.9 (2.58)
  Day 30: number analyzed (Participants) | 89
  Day 30 | 12.0 (2.50)
  Day 60: number analyzed (Participants) | 89
  Day 60 | 11.8 (2.53)
  Day 90: number analyzed (Participants) | 89
  Day 90 | 11.7 (2.73)
  Day 135: number analyzed (Participants) | 85
  Day 135 | 11.9 (2.78)
  Day 180: number analyzed (Participants) | 86
  Day 180 | 11.8 (2.57)

8. Primary Outcome: Lens Wear Time at Each Visit Day
Description: Subject recorded a response to the question, "How many hours have you worn your contact lenses today?" Lens wear was measured in hours. Habitual lenses were used at the Day 0 time point.
Time Frame: Day 0, Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set, with non-missing response
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | FID 120947A
Number analyzed (Participants) | 90
hours
  Day 0 | 4.3 (3.53)
  Day 7 | 4.8 (3.53)
  Day 30: number analyzed (Participants) | 89
  Day 30 | 4.7 (3.27)
  Day 60: number analyzed (Participants) | 89
  Day 60 | 4.2 (3.04)
  Day 90: number analyzed (Participants) | 89
  Day 90 | 4.4 (3.33)
  Day 135: number analyzed (Participants) | 85
  Day 135 | 4.4 (3.28)
  Day 180: number analyzed (Participants) | 86
  Day 180 | 4.6 (3.35)

9. Primary Outcome: Average Rewetting Drop Frequency at Each Visit
Description: Subject recorded a response to the question, "Averaging over the last 3 days, how many times per day did you use rewetting drops?" Habitual lenses were used at the Day 0 time point.
Time Frame: Day 0, Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set, with non-missing response
Measure: Mean (Standard Deviation); unit: times per day
Arm/Group | FID 120947A
Number analyzed (Participants) | 90
times per day
  Day 0 | 0.3 (1.11)
  Day 7 | 1.4 (2.27)
  Day 30: number analyzed (Participants) | 89
  Day 30 | 1.7 (1.85)
  Day 60: number analyzed (Participants) | 89
  Day 60 | 1.6 (1.79)
  Day 90: number analyzed (Participants) | 89
  Day 90 | 1.7 (1.93)
  Day 135: number analyzed (Participants) | 85
  Day 135 | 1.8 (1.97)
  Day 180: number analyzed (Participants) | 86
  Day 180 | 1.7 (2.00)

10. Primary Outcome: Number of Unscheduled Lens Replacements by Reason
Description: Subjects were dispensed enough contact lenses to follow a 2-week replacement schedule during the study. Lenses replaced at other times were considered unscheduled. The counts in the table represent the total number of unscheduled lenses replaced by reason for any eye, any subject. All lenses which were replaced are counted. Habitual lenses were used at the Day 0 time point.
Time Frame: Up to Day 180
Population: Full Analysis Set, with specified reason for replacement.
Measure: Number; unit: lenses
Arm/Group | FID 120947A
Number analyzed (Participants) | 90
lenses
  Unplanned - Lens torn on eye | 5
  Unplanned - Lens torn while handling | 38
  Unplanned - Lens deposit | 17
  Unplanned - Bad edge | 4
  Unplanned - Bad surface | 0
  Unplanned - Discoloration | 0
  Unplanned - No lens in pack | 0
  Unplanned - Visual Acuity | 2
  Unplanned - Discomfort | 6
  Unplanned - Pathology | 0
  Unplanned - Lost | 7
  Other | 2

11. Primary Outcome: Likert Item - "When I Use This Solution, my Lenses Are Comfortable All Day."
Description: Lens comfort was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects. Habitual lenses and habitual lens care solution were used at the Day 0 time point.
Time Frame: Day 0, Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | Strongly Agree | Agree | Undecided | Disagree | Strongly Disagree
Number analyzed (Participants) | 90 | 90 | 90 | 90 | 90
percentage of subjects
  Day 0 | 26.7 | 44.4 | 22.2 | 6.7 | 0.0
  Day 7 | 35.6 | 41.1 | 15.6 | 7.8 | 0.0
  Day 30: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 30 | 29.2 | 48.3 | 13.5 | 9.0 | 0.0
  Day 60: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 60 | 34.8 | 46.1 | 14.6 | 4.5 | 0.0
  Day 90: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 90 | 36.0 | 49.4 | 11.2 | 2.2 | 1.1
  Day 135: number analyzed (Participants) | 85 | 85 | 85 | 85 | 85
  Day 135 | 38.8 | 44.7 | 16.5 | 0.0 | 0.0
  Day 180: number analyzed (Participants) | 86 | 86 | 86 | 86 | 86
  Day 180 | 41.9 | 50.0 | 8.1 | 0.0 | 0.0

12. Primary Outcome: Likert Item - "When I Use This Solution, at the End of the Lens Wearing Day my Vision is Clear."
Description: Clear vision was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects. Habitual lenses and habitual lens care solution were used at the Day 0 time point.
Time Frame: Day 0, Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set with non-missing response
Measure: Number; unit: percentage of subjects
Arm/Group | Strongly Agree | Agree | Undecided | Disagree | Strongly Disagree
Number analyzed (Participants) | 90 | 90 | 90 | 90 | 90
percentage of subjects
  Day 0 | 42.2 | 38.9 | 12.2 | 5.6 | 1.1
  Day 7 | 48.9 | 37.8 | 10.0 | 3.3 | 0.0
  Day 30: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 30 | 46.1 | 37.1 | 14.6 | 2.2 | 0.0
  Day 60: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 60 | 42.7 | 41.6 | 13.5 | 2.2 | 0.0
  Day 90: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 90 | 39.3 | 47.2 | 13.5 | 0.0 | 0.0
  Day 135: number analyzed (Participants) | 85 | 85 | 85 | 85 | 85
  Day 135 | 41.2 | 47.1 | 10.6 | 0.0 | 1.2
  Day 180: number analyzed (Participants) | 86 | 86 | 86 | 86 | 86
  Day 180 | 44.2 | 48.8 | 7.0 | 0.0 | 0.0

13. Primary Outcome: Likert Item - "When I Use This Solution, I Like the Way This Product Feels During Handling."
Description: Product handling was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects. Habitual lenses and habitual lens care solution were used at the Day 0 time point.
Time Frame: Day 0, Day 7, Day 30, Day 60, Day 90, Day 135, Day 180
Population: Full Analysis Set with non-missing response
Measure: Number; unit: percentage of subjects
Arm/Group | Strongly Agree | Agree | Undecided | Disagree | Strongly Disagree
Number analyzed (Participants) | 90 | 90 | 90 | 90 | 90
percentage of subjects
  Day 0 | 44.4 | 41.1 | 12.2 | 2.2 | 0.0
  Day 7 | 28.9 | 32.2 | 25.6 | 12.2 | 1.1
  Day 30: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 30 | 31.5 | 39.3 | 19.1 | 7.9 | 2.2
  Day 60: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 60 | 25.8 | 40.4 | 27.0 | 5.6 | 1.1
  Day 90: number analyzed (Participants) | 89 | 89 | 89 | 89 | 89
  Day 90 | 30.3 | 41.6 | 22.5 | 3.4 | 2.2
  Day 135: number analyzed (Participants) | 85 | 85 | 85 | 85 | 85
  Day 135 | 29.4 | 44.7 | 21.2 | 2.4 | 2.4
  Day 180: number analyzed (Participants) | 86 | 86 | 86 | 86 | 86
  Day 180 | 34.9 | 40.7 | 19.8 | 2.3 | 2.3

ADVERSE EVENTS:
Time Frame: Day 1 through study completion, an average of 6 months
Description: An AE was defined as any unfavorable or unintended sign, symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. "At Risk" population for ocular AEs is included with unit of "eyes."
Groups:
- FID 120977A - Subject Based Adverse Events: All subjects treated with FID 120947A contact lens disinfecting solution
- FID 120977A - Ocular Adverse Events: All eyes treated with FID 120947A contact lens disinfecting solution
Arm/Group | FID 120977A - Subject Based Adverse Events | FID 120977A - Ocular Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/180
Other Adverse Events (participants affected / at risk) | 0/90 | 25/180
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FID 120977A - Subject Based Adverse Events (N=90) | FID 120977A - Ocular Adverse Events (N=180)
Eye irritation (Eye disorders) | 0 | 11
Vision blurred (Eye disorders) | 0 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.